CLINICAL TRIAL: NCT01947621
Title: International Multicenter Registry on Takotsubo Cardiomyopathy
Brief Title: International Takotsubo Registry (InterTAK Registry)
Acronym: InterTAK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Collaborators: University of California, Davis (Other); Hannover Medical School (Other); Ludwig-Maximilians - University of Munich (Other); University of Heidelberg Medical Center (Other); University Hospital Schleswig-Holstein (Other); Charite University, Berlin, Germany (Other); University of Kentucky (Other); Medical University of Cologne (Other); University Hospital, Saarland (Other); University Hospital, Essen (Other); Asklepios Kliniken Hamburg GmbH (Other); University Hospital Goettingen (Other); University of Magdeburg (Other); Oxford University Hospitals NHS Trust (Other); Kantonsspital Winterthur KSW (Other); Turku University Hospital (Other Government); Medical University of Gdansk (Other); Medical University of Warsaw (Other); University Hospital, Basel, Switzerland (Other); Catholic University of the Sacred Heart (Other); Medical University Innsbruck (Other); Cardiocentro Ticino (Other); Luzerner Kantonsspital (Other); Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: InterTAK Registry
Record Dates: First submitted 2013-09-09; First posted 2013-09-20 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Takotsubo Cardiomyopathy
Keywords: Broken heart syndrome, stress cardiomyopathy
MeSH Terms: conditions — Takotsubo Cardiomyopathy

STUDY DESIGN:
Observational Model: Cohort

INTERVENTIONS:
Other:

SUMMARY:
This is a multicenter, multinational, prospective and retrospective, observational study of patients with Takotsubo cardiomyopathy (TTC).

Data on natural profile (demographical characteristics, clinical phenotype, laboratory values, electrocardiography parameters, echocardiography parameters, coronary angiography parameters, medication) and outcome are systematically collected.

Our aim is to gain a better insight into the clinical profile and pathophysiology of TTC.

DETAILED DESCRIPTION:
Registry is an open-ended study and eligible individuals are assessed at index event and follow-up on their phenotypical characteristics. Furthermore, outcome data are collected (by clinical visits or telephone follow-up).

In addition, participants are given the option to consent to the donation of biosamples for the purposes to identify TTC specific biomarkers and mutations (sub-study on behalf of the registry).

ELIGIBILITY:
Inclusion criteria: Mayo Clinic Diagnostic Criteria (Prasad et al. American Heart Journal 2008)

1. Transient hypokinesis, akinesis, or dyskinesis of the left ventricular mid segments with or without apical involvement; the regional wall motion abnormalities extend beyond a single epicardial vascular distribution; a stressful trigger is often, but not always present.*
2. Absence of obstructive coronary disease or angiographic evidence of acute plaque rupture. †
3. New electrocardiographic abnormalities (either ST-segment elevation and/or T-wave inversion) or modest elevation in cardiac troponin.

In both of the above circumstances, the diagnosis of TTC should be made with caution, and a clear stressful precipitating trigger must be sought. * There are rare exceptions to these criteria such as those patients in whom the regional wall motion abnormality is limited to a single coronary territory.

† It is possible that a patient with obstructive coronary atherosclerosis may also develop TTC.

Exclusion criteria: Patients with Myocarditis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with manifest Takotsubo cardiomyopathy
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2011-01; Primary Completion 2014-10 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Natural history of TTC | 10 years
  To determine the natural history of Takotsubo cardiomyopathy.

SECONDARY OUTCOMES:
Cardiovascular complications, recurrence of TTC and all cause mortality | at hospitalizsation, short term (1 year) and long term (10 years)
  Patients will be assessed for cardiovascular complications during hospitalisation and at follow-up (up to 10 years)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Templin, MD, PhD, Principal Investigator — University Hospital Zurich, Division of Cardiology
Locations (1):
- University Hospital Zurich, Division of Cardiology, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Stahli B, Schweiger V, Cammann VL, Schindler M, Szawan KA, Niederseer D, Wurdinger M, Schonberger A, Schonberger M, Koleva I, Mercier JC, Petkova V, Steigmeier M, Citro R, Bossone E, Luscher TF, Templin-Ghadri JR, Di Vece D, Templin C; InterTAK Collaborators. Body weight and mortality in Takotsubo syndrome: insights from the International Takotsubo (InterTAK) Registry. Open Heart. 2026 Jan 29;13(1):e003851. doi: 10.1136/openhrt-2025-003851. PMID 41611312
- [Derived] Cammann VL, Scheitz JF, von Rennenberg R, Jancke L, Nolte CH, Szawan KA, Stengl H, Wurdinger M, Endres M, Templin C, Ghadri JR; InterTAK Consortium. Clinical correlates and prognostic impact of neurologic disorders in Takotsubo syndrome. Sci Rep. 2021 Dec 7;11(1):23555. doi: 10.1038/s41598-021-01496-9. PMID 34876622
- [Derived] El-Battrawy I, Cammann VL, Kato K, Szawan KA, Di Vece D, Rossi A, Wischnewsky M, Hermes-Laufer J, Gili S, Citro R, Bossone E, Neuhaus M, Franke J, Meder B, Jaguszewski M, Noutsias M, Knorr M, Heiner S, D'Ascenzo F, Dichtl W, Burgdorf C, Kherad B, Tschope C, Sarcon A, Shinbane J, Rajan L, Michels G, Pfister R, Cuneo A, Jacobshagen C, Karakas M, Koenig W, Pott A, Meyer P, David Arroja J, Banning A, Cuculi F, Kobza R, Fischer TA, Vasankari T, Airaksinen KEJ, Napp LC, Budnik M, Dworakowski R, MacCarthy P, Kaiser C, Osswald S, Galiuto L, Chan C, Bridgman P, Beug D, Delmas C, Lairez O, Gilyarova E, Shilova A, Gilyarov M, Kozel M, Tousek P, Winchester DE, Galuszka J, Ukena C, Poglajen G, Carrilho-Ferreira P, Hauck C, Paolini C, Bilato C, Kobayashi Y, Prasad A, Rihal CS, Liu K, Schulze PC, Bianco M, Jorg L, Rickli H, Pestana G, Nguyen TH, Bohm M, Maier LS, Pinto FJ, Widimsky P, Felix SB, Opolski G, Braun-Dullaeus RC, Rottbauer W, Hasenfuss G, Pieske BM, Schunkert H, Thiele H, Bauersachs J, Katus HA, Horowitz JD, Di Mario C, Munzel T, Crea F, Bax JJ, Luscher TF, Ruschitzka F, Duru F, Borggrefe M, Ghadri JR, Akin I, Templin C. Impact of Atrial Fibrillation on Outcome in Takotsubo Syndrome: Data From the International Takotsubo Registry. J Am Heart Assoc. 2021 Aug 3;10(15):e014059. doi: 10.1161/JAHA.119.014059. Epub 2021 Jul 28. PMID 34315238
- [Derived] Cammann VL, Sarcon A, Szawan KA, Wurdinger M, Azam S, Shinbane J, Seifert B, Ghadri JR, Saw J, Templin C. Clinical characteristics and outcomes of patients with takotsubo syndrome versus spontaneous coronary artery dissection. Cardiol J. 2023;30(1):125-130. doi: 10.5603/CJ.a2021.0065. Epub 2021 Jun 24. PMID 34165180
- [Derived] Imori Y, Kato K, Cammann VL, Szawan KA, Wischnewsky M, Dreiding S, Wurdinger M, Schonberger M, Petkova V, Niederseer D, Levinson RA, Di Vece D, Gili S, Seifert B, Wakita M, Suzuki N, Citro R, Bossone E, Heiner S, Knorr M, Jansen T, Munzel T, D'Ascenzo F, Franke J, Sorici-Barb I, Katus HA, Sarcon A, Shinbane J, Napp LC, Bauersachs J, Jaguszewski M, Shiomura R, Nakamura S, Takano H, Noutsias M, Burgdorf C, Ishibashi I, Himi T, Koenig W, Schunkert H, Thiele H, Kherad B, Tschope C, Pieske BM, Rajan L, Michels G, Pfister R, Mizuno S, Cuneo A, Jacobshagen C, Hasenfuss G, Karakas M, Mochizuki H, Pott A, Rottbauer W, Said SM, Braun-Dullaeus RC, Banning A, Isogai T, Kimura A, Cuculi F, Kobza R, Fischer TA, Vasankari T, Airaksinen KEJ, Tomita Y, Budnik M, Opolski G, Dworakowski R, MacCarthy P, Kaiser C, Osswald S, Galiuto L, Crea F, Dichtl W, Murakami T, Ikari Y, Empen K, Beug D, Felix SB, Delmas C, Lairez O, Yamaguchi T, El-Battrawy I, Akin I, Borggrefe M, Horowitz JD, Kozel M, Tousek P, Widimsky P, Gilyarova E, Shilova A, Gilyarov M, Neuhaus M, Meyer P, Arroja JD, Chan C, Bridgman P, Galuszka J, Poglajen G, Carrilho-Ferreira P, Pinto FJ, Hauck C, Maier LS, Liu K, Di Mario C, Paolini C, Bilato C, Bianco M, Jorg L, Rickli H, Winchester DE, Ukena C, Bohm M, Bax JJ, Prasad A, Rihal CS, Saito S, Kobayashi Y, Luscher TF, Ruschitzka F, Shimizu W, Ghadri JR, Templin C. Ethnic comparison in takotsubo syndrome: novel insights from the International Takotsubo Registry. Clin Res Cardiol. 2022 Feb;111(2):186-196. doi: 10.1007/s00392-021-01857-4. Epub 2021 May 19. PMID 34013386
- [Derived] Napp LC, Cammann VL, Jaguszewski M, Szawan KA, Wischnewsky M, Gili S, Knorr M, Heiner S, Citro R, Bossone E, D'Ascenzo F, Neuhaus M, Franke J, Sorici-Barb I, Noutsias M, Burgdorf C, Koenig W, Kherad B, Sarcon A, Rajan L, Michels G, Pfister R, Cuneo A, Jacobshagen C, Karakas M, Pott A, Meyer P, Arroja JD, Banning A, Cuculi F, Kobza R, Fischer TA, Vasankari T, Airaksinen KEJ, Hauck C, Paolini C, Bilato C, Imori Y, Kato K, Kobayashi Y, Opolski G, Budnik M, Dworakowski R, MacCarthy P, Kaiser C, Osswald S, Galiuto L, Dichtl W, Chan C, Bridgman P, Beug D, Delmas C, Lairez O, El-Battrawy I, Akin I, Gilyarova E, Shilova A, Gilyarov M, Horowitz JD, Polednikova K, Tousek P, Widimsky P, Winchester DE, Galuszka J, Ukena C, Poglajen G, Carrilho-Ferreira P, Di Mario C, Prasad A, Rihal CS, Schulze PC, Bianco M, Crea F, Borggrefe M, Maier LS, Pinto FJ, Braun-Dullaeus RC, Rottbauer W, Katus HA, Hasenfuss G, Tschope C, Pieske BM, Thiele H, Schunkert H, Bohm M, Felix SB, Munzel T, Bax JJ, Bauersachs J, Braunwald E, Luscher TF, Ruschitzka F, Ghadri JR, Templin C. Coexistence and outcome of coronary artery disease in Takotsubo syndrome. Eur Heart J. 2020 Sep 7;41(34):3255-3268. doi: 10.1093/eurheartj/ehaa210. PMID 32484517
- [Derived] D'Ascenzo F, Gili S, Bertaina M, Iannaccone M, Cammann VL, Di Vece D, Kato K, Saglietto A, Szawan KA, Frangieh AH, Boffini B, Annaratone M, Sarcon A, Levinson RA, Franke J, Napp LC, Jaguszewski M, Noutsias M, Munzel T, Knorr M, Heiner S, Katus HA, Burgdorf C, Schunkert H, Thiele H, Bauersachs J, Tschope C, Pieske BM, Rajan L, Michels G, Pfister R, Cuneo A, Jacobshagen C, Hasenfuss G, Karakas M, Koenig W, Rottbauer W, Said SM, Braun-Dullaeus RC, Banning A, Cuculi F, Kobza R, Fischer TA, Vasankari T, Airaksinen KEJ, Opolski G, Dworakowski R, MacCarthy P, Kaiser C, Osswald S, Galiuto L, Crea F, Dichtl W, Franz WM, Empen K, Felix SB, Delmas C, Lairez O, El-Battrawy I, Akin I, Borggrefe M, Horowitz JD, Kozel M, Tousek P, Widimsky P, Gilyarova E, Shilova A, Gilyarov M, Biondi-Zoccai G, Winchester DE, Ukena C, Neuhaus M, Bax JJ, Prasad A, Di Mario C, Bohm M, Gasparini M, Ruschitzka F, Bossone E, Citro R, Rinaldi M, De Ferrari GM, Luscher T, Ghadri JR, Templin C. Impact of aspirin on takotsubo syndrome: a propensity score-based analysis of the InterTAK Registry. Eur J Heart Fail. 2020 Feb;22(2):330-337. doi: 10.1002/ejhf.1698. Epub 2019 Dec 20. PMID 31863563
- [Derived] Ding KJ, Cammann VL, Szawan KA, Stahli BE, Wischnewsky M, Di Vece D, Citro R, Jaguszewski M, Seifert B, Sarcon A, Knorr M, Heiner S, Gili S, D'Ascenzo F, Neuhaus M, Napp LC, Franke J, Noutsias M, Burgdorf C, Koenig W, Kherad B, Rajan L, Michels G, Pfister R, Cuneo A, Jacobshagen C, Karakas M, Pott A, Meyer P, Arroja JD, Banning A, Cuculi F, Kobza R, Fischer TA, Vasankari T, Airaksinen KEJ, Paolini C, Bilato C, Carrilho-Ferreira P, Opolski G, Dworakowski R, MacCarthy P, Kaiser C, Osswald S, Galiuto L, Dichtl W, Chan C, Bridgman P, Delmas C, Lairez O, El-Battrawy I, Akin I, Gilyarova E, Shilova A, Gilyarov M, Kozel M, Tousek P, Widimsky P, Winchester DE, Galuszka J, Ukena C, Horowitz JD, Di Mario C, Prasad A, Rihal CS, Pinto FJ, Crea F, Borggrefe M, Braun-Dullaeus RC, Rottbauer W, Bauersachs J, Katus HA, Hasenfuss G, Tschope C, Pieske BM, Thiele H, Schunkert H, Bohm M, Felix SB, Munzel T, Bax JJ, Luscher TF, Ruschitzka F, Ghadri JR, Bossone E, Templin C. Intraventricular Thrombus Formation and Embolism in Takotsubo Syndrome: Insights From the International Takotsubo Registry. Arterioscler Thromb Vasc Biol. 2020 Jan;40(1):279-287. doi: 10.1161/ATVBAHA.119.313491. Epub 2019 Nov 26. PMID 31766870
- [Derived] Jurisic S, Gili S, Cammann VL, Kato K, Szawan KA, D'Ascenzo F, Jaguszewski M, Bossone E, Citro R, Sarcon A, Napp LC, Franke J, Noutsias M, Knorr M, Heiner S, Burgdorf C, Koenig W, Pott A, Kherad B, Rajan L, Michels G, Pfister R, Cuneo A, Jacobshagen C, Karakas M, Meyer P, Arroja JD, Banning A, Cuculi F, Kobza R, Fischer TA, Vasankari T, Airaksinen KEJ, Dworakowski R, Kaiser C, Osswald S, Galiuto L, Dichtl W, Chan C, Bridgman P, Beug D, Delmas C, Lairez O, Kozel M, Tousek P, Winchester DE, Gilyarova E, Shilova A, Gilyarov M, El-Battrawy I, Akin I, Galuszka J, Ukena C, Poglajen G, Paolini C, Bilato C, Carrilho-Ferreira P, Pinto FJ, Opolski G, MacCarthy P, Kobayashi Y, Prasad A, Rihal CS, Widimsky P, Horowitz JD, Di Mario C, Crea F, Tschope C, Pieske BM, Hasenfuss G, Rottbauer W, Braun-Dullaeus RC, Felix SB, Borggrefe M, Thiele H, Bauersachs J, Katus HA, Schunkert H, Munzel T, Bohm M, Bax JJ, Luscher TF, Ruschitzka F, Ghadri JR, Templin C. Clinical Predictors and Prognostic Impact of Recovery of Wall Motion Abnormalities in Takotsubo Syndrome: Results From the International Takotsubo Registry. J Am Heart Assoc. 2019 Nov 5;8(21):e011194. doi: 10.1161/JAHA.118.011194. Epub 2019 Nov 1. PMID 31672100
- [Derived] Cammann VL, Sarcon A, Ding KJ, Seifert B, Kato K, Di Vece D, Szawan KA, Gili S, Jurisic S, Bacchi B, Micek J, Frangieh AH, Napp LC, Jaguszewski M, Bossone E, Citro R, D'Ascenzo F, Franke J, Noutsias M, Knorr M, Heiner S, Burgdorf C, Koenig W, Thiele H, Tschope C, Rajan L, Michels G, Pfister R, Cuneo A, Jacobshagen C, Karakas M, Banning A, Cuculi F, Kobza R, Fischer TA, Vasankari T, Airaksinen KEJ, Dworakowski R, Kaiser C, Osswald S, Galiuto L, Dichtl W, Delmas C, Lairez O, Horowitz JD, Kozel M, Widimsky P, Tousek P, Winchester DE, Gilyarova E, Shilova A, Gilyarov M, El-Battrawy I, Akin I, Ukena C, Bauersachs J, Pieske BM, Hasenfuss G, Rottbauer W, Braun-Dullaeus RC, Opolski G, MacCarthy P, Felix SB, Borggrefe M, Di Mario C, Crea F, Katus HA, Schunkert H, Munzel T, Bohm M, Bax JJ, Prasad A, Shinbane J, Luscher TF, Ruschitzka F, Ghadri JR, Templin C. Clinical Features and Outcomes of Patients With Malignancy and Takotsubo Syndrome: Observations From the International Takotsubo Registry. J Am Heart Assoc. 2019 Aug 6;8(15):e010881. doi: 10.1161/JAHA.118.010881. Epub 2019 Jul 17. PMID 31311438
- [Derived] Kato K, Di Vece D, Cammann VL, Micek J, Szawan KA, Bacchi B, Luscher TF, Ruschitzka F, Ghadri JR, Templin C; InterTAK Collaborators. Takotsubo Recurrence: Morphological Types and Triggers and Identification of Risk Factors. J Am Coll Cardiol. 2019 Mar 5;73(8):982-984. doi: 10.1016/j.jacc.2018.12.033. No abstract available. PMID 30819368
- [Derived] Ghadri JR, Kato K, Cammann VL, Gili S, Jurisic S, Di Vece D, Candreva A, Ding KJ, Micek J, Szawan KA, Bacchi B, Bianchi R, Levinson RA, Wischnewsky M, Seifert B, Schlossbauer SA, Citro R, Bossone E, Munzel T, Knorr M, Heiner S, D'Ascenzo F, Franke J, Sarcon A, Napp LC, Jaguszewski M, Noutsias M, Katus HA, Burgdorf C, Schunkert H, Thiele H, Bauersachs J, Tschope C, Pieske BM, Rajan L, Michels G, Pfister R, Cuneo A, Jacobshagen C, Hasenfuss G, Karakas M, Koenig W, Rottbauer W, Said SM, Braun-Dullaeus RC, Banning A, Cuculi F, Kobza R, Fischer TA, Vasankari T, Airaksinen KEJ, Opolski G, Dworakowski R, MacCarthy P, Kaiser C, Osswald S, Galiuto L, Crea F, Dichtl W, Empen K, Felix SB, Delmas C, Lairez O, El-Battrawy I, Akin I, Borggrefe M, Horowitz J, Kozel M, Tousek P, Widimsky P, Gilyarova E, Shilova A, Gilyarov M, Winchester DE, Ukena C, Bax JJ, Prasad A, Bohm M, Luscher TF, Ruschitzka F, Templin C. Long-Term Prognosis of Patients With Takotsubo Syndrome. J Am Coll Cardiol. 2018 Aug 21;72(8):874-882. doi: 10.1016/j.jacc.2018.06.016. PMID 30115226
- [Derived] Bohm M, Cammann VL, Ghadri JR, Ukena C, Gili S, Di Vece D, Kato K, Ding KJ, Szawan KA, Micek J, Jurisic S, D'Ascenzo F, Frangieh AH, Rechsteiner D, Seifert B, Ruschitzka F, Luscher T, Templin C; InterTAK Collaborators. Interaction of systolic blood pressure and resting heart rate with clinical outcomes in takotsubo syndrome: insights from the International Takotsubo Registry. Eur J Heart Fail. 2018 Jun;20(6):1021-1030. doi: 10.1002/ejhf.1162. Epub 2018 Mar 8. PMID 29517122
- [Derived] Borchert T, Hubscher D, Guessoum CI, Lam TD, Ghadri JR, Schellinger IN, Tiburcy M, Liaw NY, Li Y, Haas J, Sossalla S, Huber MA, Cyganek L, Jacobshagen C, Dressel R, Raaz U, Nikolaev VO, Guan K, Thiele H, Meder B, Wollnik B, Zimmermann WH, Luscher TF, Hasenfuss G, Templin C, Streckfuss-Bomeke K. Catecholamine-Dependent beta-Adrenergic Signaling in a Pluripotent Stem Cell Model of Takotsubo Cardiomyopathy. J Am Coll Cardiol. 2017 Aug 22;70(8):975-991. doi: 10.1016/j.jacc.2017.06.061. PMID 28818208
- [Derived] Ghadri JR, Cammann VL, Jurisic S, Seifert B, Napp LC, Diekmann J, Bataiosu DR, D'Ascenzo F, Ding KJ, Sarcon A, Kazemian E, Birri T, Ruschitzka F, Luscher TF, Templin C; InterTAK co-investigators. A novel clinical score (InterTAK Diagnostic Score) to differentiate takotsubo syndrome from acute coronary syndrome: results from the International Takotsubo Registry. Eur J Heart Fail. 2017 Aug;19(8):1036-1042. doi: 10.1002/ejhf.683. Epub 2016 Dec 7. PMID 27928880
- [Derived] Frangieh AH, Obeid S, Ghadri JR, Imori Y, D'Ascenzo F, Kovac M, Ruschitzka F, Luscher TF, Duru F, Templin C; InterTAK Collaborators. ECG Criteria to Differentiate Between Takotsubo (Stress) Cardiomyopathy and Myocardial Infarction. J Am Heart Assoc. 2016 Jun 13;5(6):e003418. doi: 10.1161/JAHA.116.003418. PMID 27412903
- [Derived] Templin C, Ghadri JR, Diekmann J, Napp LC, Bataiosu DR, Jaguszewski M, Cammann VL, Sarcon A, Geyer V, Neumann CA, Seifert B, Hellermann J, Schwyzer M, Eisenhardt K, Jenewein J, Franke J, Katus HA, Burgdorf C, Schunkert H, Moeller C, Thiele H, Bauersachs J, Tschope C, Schultheiss HP, Laney CA, Rajan L, Michels G, Pfister R, Ukena C, Bohm M, Erbel R, Cuneo A, Kuck KH, Jacobshagen C, Hasenfuss G, Karakas M, Koenig W, Rottbauer W, Said SM, Braun-Dullaeus RC, Cuculi F, Banning A, Fischer TA, Vasankari T, Airaksinen KE, Fijalkowski M, Rynkiewicz A, Pawlak M, Opolski G, Dworakowski R, MacCarthy P, Kaiser C, Osswald S, Galiuto L, Crea F, Dichtl W, Franz WM, Empen K, Felix SB, Delmas C, Lairez O, Erne P, Bax JJ, Ford I, Ruschitzka F, Prasad A, Luscher TF. Clinical Features and Outcomes of Takotsubo (Stress) Cardiomyopathy. N Engl J Med. 2015 Sep 3;373(10):929-38. doi: 10.1056/NEJMoa1406761. PMID 26332547
- See also: Related Info — http://www.takotsubo-registry.com